CLINICAL TRIAL: NCT02560870
Title: Randomized, Clinical Trial to Evaluate the Effects of Aloe Vera Mouthwash in Comparison With Non-alcoholic Chlorhexidine on Periodontal Disease
Brief Title: Compare the Efficacy of Aloe Vera Mouthwash With Non- Alcoholic Chlorhexidine Mouthwash on Periodontal Diseases
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Amirhossein Farahmand, Evaluate and compare the efficacy of aloe Vera mouthwash with non- alcoholic Chlorhexidine mouthwash on periodontal diseases., Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 487
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aloe Vera mouthwash (Active Comparator): mouthwash (Aleo Vera)10 ml by patients routinely washed two times in one day for about 30 seconds for two weeks.
  Interventions: Drug: Active Comparator:Aloe Vera mouthwash
- Chlorhexidine mouthwash (Active Comparator): mouthwash (Chlorhexidine )10 ml by patients routinely washed two times in one day for about 30 seconds for two weeks.
  Interventions: Drug: Active Comparator:Chlorhexidine mouthwash

INTERVENTIONS:
Drug: Active Comparator:Aloe Vera mouthwash — mouthwash( Aloe Vera),10 ml by patients routinely washed two times in one day for about 30 seconds for two weeks.
  Other Names: Aloe Vera mouthwash made by Alodent Co. UK
  Arms: Aloe Vera mouthwash
Drug: Active Comparator:Chlorhexidine mouthwash — mouthwash( Chlorhexidine ),10 ml by patients routinely washed two times in one day for about 30 seconds for two weeks.
  Other Names: Chlorhexidine mouthwash made by Perio-Kin, Livar CO. Spain
  Arms: Chlorhexidine mouthwash

SUMMARY:
Aim: To compare the efficacy of Aloe Vera and non-alcoholic chlorhexidine mouthwash in the treatment of Periodontal diseases.

Methods &Material: 32 patients were selected, the following periodontal parameters were recorded at baseline, and after recording all the parameters at the baseline, Scaling, root planning, and polishing are done for all the patients participating in the study. Oral hygiene instructions were given that included brushing twice a day with a soft brush, After 2 weeks, patients in the study, were randomly (Balanced Block Randomization) equal divided into 2 groups;

Group A: mouthwash aloe Vera (Alodent Co. UK) for each patient, Group B: Non-alcoholic Chlorhexidine (Perio-Kin, Livar CO. Spain) 10 ml by patients routinely washed two times in one day for about 30 seconds and lasts for 15 days, then every 7 days periodontal parameters, and at the end of 2 weeks (days 0, 7, 15) clinical changes are evaluated.

DETAILED DESCRIPTION:
Eligible participants were 32 adult patients treated for chronic periodontitis and participating in a supportive periodontal therapy program at the Department of Periodontology of the Dental Clinic of the Islamic Azad University, Dental Branch of Tehran were included in the current study; Recruitment of participants started july 2014 and ended may 2015. The study met the criteria of the Helsinki Declaration of 1975, revised in 2008. The survey plan was reviewed and sanctioned, approved by the ethics commission of the Institutional Ethical Committee and Review Board of the Deputy of Research, School of Dentistry. All subjects received the oral and written explanation of the intent of the survey and signed an informed consent after receiving detailed information about the purpose, the benefits, and the possible risks associated with the trial. Individuals satisfying the following entry criteria were recruited:

* Diagnosed suffering from initial (early) to moderate chronic periodontitis;
* Adult patients, more than 28 years old with at least 20 remaining teeth and at least three teeth in each quadrant;
* The presence of at least two residual sites with a probing pocket depth (PPD>4 mm in two opposite quadrants, which showed bleeding upon probing, radiographically comparable amount of periodontal breakdown and good matching in tooth type, also clinical and minimal radiographic signs of initial (early) to moderate (clinical attachment level of 1 to 3mm.

ELIGIBILITY:
Inclusion Criteria:

* Presence of two periodontal sites located on the same side pocket depth 4 mm or more.
* Chronic periodontitis patients.

Exclusion Criteria:

* Orthodontic treatment.
* Use removal denture.
* Presence of vertical bone defect.
* Use of medicine therapy within the 3 months prior to the study.
* Allergy to chlorhexidine and Aloe Vera.
* smoking.
* Systemic diseases that could influence the course of periodontal disease.
* Pregnancy and lactation.
* Aggressive periodontitis.
* Furcation involvement.
* Periodontal therapy 6 months prior to the study.
* Extensive caries.

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Reduction of pocket depth | 7days
  Periodontal pobe

SECONDARY OUTCOMES:
Reduction of bleeding on probing | 7days
  Periodontal pobe
Reduction of plaque index | 7days
  Plaque Index(O'Leary )